CLINICAL TRIAL: NCT05465941
Title: Phase II Clinical Trial of PLX038 in Patients With Platinum-Resistant Ovarian, Primary Peritoneal, and Fallopian Tube Cancer
Brief Title: PLX038 for Treatment of Metastatic Platinum-resistant Ovarian, Primary Peritoneal, and Fallopian Tube Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC210601; P50CA136393 (NIH); NCI-2022-04925 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-012233 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Biopsy; Specimen Handling

STUDY DESIGN:
Masking Description: Staining will be read independently by two individuals blinded to treatment, who will score each sample for the percentage of cells that are positive for >8 nucleoplasmic TOP1ccs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pegylated SN-38 conjugate PLX038) (Experimental): Patients receive PLX038 IV over 1 hour on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, biopsy, as well as blood and stool sample collection during screening and on the trial.
  Interventions: Procedure: Biopsy; Drug: Pegylated SN-38 Conjugate PLX038; Procedure: Computed Tomography; Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: Bx; BIOPSY_TYPE
Drug: Pegylated SN-38 Conjugate PLX038 — Given IV
  Other Names: Pegylated SN-38 PLX038; PLX 038; PLX-038; PLX038
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT SCAN; tomography
Procedure: Biospecimen Collection — Undergo blood and stool sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase II trial tests whether pegylated SN-38 conjugate PLX038 (PLX038) works to shrink tumors in patients with ovarian, primary peritoneal, and fallopian tube cancers that has spread from where it first started (primary site) to other places in the body (metastatic). PLX038 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the overall tumor response rate (overall response rate [ORR], that is, complete response [CR] + partial response [PR], according to Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1] of PLX038 in the setting of metastatic platinum resistant high grade serous ovarian cancer.

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival and overall survival of treatment with PLX038.

II. To describe and assess tolerability of PLX038. III. Measure PLX038 induced tumor TOP1-deoxyribonucleic acid (DNA) covalent complexes (TOP1cc) in pretreatment and Cycle 1 Day 8 biopsies to confirm persistent stabilization of TOP1cc and evaluate association with tumor response rate.

CORRELATIVE RESEARCH:

I. Measure TOP1cc in circulating tumor cells and evaluate association with TOP1cc in tumor tissue and tumor response rate.

II. Assess homologous repair status and association with tumor response. III. Assess expression of SN-38 transports by quantitative reverse transcriptase-polymerase chain reaction (RT-PCR) and association with tumor response.

IV. Assess pharmacokinetics of SN-38 and SN-38G as well as their association with gastrointestinal (GI) toxicity.

V. Assess the gut microbiota and evaluate association with GI toxicity profile.

OUTLINE:

Patients receive PLX038 intravenously (IV) over 1 hour on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT), biopsy, as well as blood and stool sample collection during screening and on the trial.

After completion of study treatment, patients are followed up at 30 days and every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years NOTE: Because no dosing or adverse event data are currently available on the use of PLX038 in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Histological confirmed high grade serous ovarian cancer consistent with ovarian, fallopian tube, or primary peritoneal carcinoma (NOTE: Any of these diseases are referred to in this protocol as "ovarian cancer")
* Recurrent high grade serous ovarian cancer that was initially platinum sensitive (i.e., had at least one platinum-free interval of at least 6 months before progression) is now platinum resistant
* No more than one prior line of therapy for platinum resistant disease. NOTE: Prior poly adenosine diphosphate-ribose polymerase (PARP) inhibitor therapy is allowed
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Disease that is amenable to two biopsies
* Life expectancy greater >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Hemoglobin >= 8.0 g/dL (obtained =< 28 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 28 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 28 days prior to registration)
* Total bilirubin >= 1.5 x upper limit of normal (ULN) (obtained =< 28 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =< 28 days prior to registration)
* Calculated creatinine clearance >= 45 ml/min using the Cockcroft-Gault formula (obtained =< 28 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research

Exclusion Criteria:

* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Histology other than high grade serous carcinoma
* Prior treatment restrictions

  * Chemotherapy =< 4 weeks prior to registration
  * Immunotherapy =< 4 weeks prior to registration
  * Radiotherapy =< 4 weeks prior to registration
  * Any other investigational therapy =< 4 weeks prior to registration
* History of prior or concurrent malignancy =< 2 years prior to registration

  * Exceptions: If natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Uncontrolled intercurrent illness including, but not limited to:

  * Myocardial infarction within 6 months of study entry
  * New York Heart Association (NYHA) class III or IV heart failure
  * Uncontrolled dysrhythmias or poorly controlled angina
  * History of serious ventricular arrhythmia (ventricular tachycardia [VT] or ventricular fibrillation [VF]) and/or factors that predispose to arrhythmia (e.g., heart failure, hypokalemia, family history of long QT syndrome)
* Known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, Exception: Patients should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this trial, patients should be class IIB or better Exception: Patients who have received prior doxorubicin (Doxil) are eligible if asymptomatic with QTc =< 480msec (Fridericia) and NYHA class IIB or better
* Known human immunodeficiency virus (HIV) Exception: Patients on effective anti-retroviral therapy with undetectable viral load =< 6 months prior to registration are eligible for this trial
* Known hepatitis

  * Exception: For patients with evidence of chronic hepatitis B virus infection the HepB viral load must be undetectable on suppressive therapy, if indicated, to be eligible
  * Exception: Patients with a history of hepatitis C virus infection must have been treated and cured. Patients with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load
* Receiving any other investigational agent
* History of clinically significant gastrointestinal bleeding, colitis, or gastrointestinal perforation
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Requirement for anticoagulation treatment that increases international normalized ratio (INR) or activated partial thromboplastin time (APTT) above the normal range (Exceptions: low dose deep vein thrombosis [DVT] or line prophylaxis allowed)
* Known central nervous system (CNS) disease Exception: Patients with treated brain metastases are eligible if follow-up brain imaging after CNS directed therapy shows no evidence of progression. Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determined that immediate CNS specific treatment is not required and is unlikely to be required during the 1st cycle of therapy
* Known Gilbert's syndrome or homozygous for the UGT1A1*28 variant allele or other relevant alleles with severely reduced UGT1A1 activity
* Patients who require treatment with UGT1A1 inhibitors during the planned period of investigational treatment with PLX038

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of confirmed tumor responses | Up to first 6 cycles of treatment (1 cycle = 21 days)
  A confirmed tumor response is defined to be either a complete response or partial response noted as the objective status on 2 consecutive evaluations at least 4 weeks apart. Confirmed tumor response will be evaluated using the first 6 cycles of treatment. All patients meeting the eligibility criteria who have signed a consent form, have begun treatment, and who have had at least one post-baseline tumor assessment will be evaluable for response. Patients not having met the criteria of having one post-baseline tumor assessment will be considered evaluable if they have discontinued the study due to disease progression.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From study entry to the first of either disease progression or death from any cause, assessed up to 5 years
  PFS will be estimated using the Kaplan-Meier method.
Overall survival (OS) | From study entry to death from any cause, assessed up to 5 years
  OS will be estimated using the Kaplan-Meier method.
Incidence of adverse event rates | Up to 30 days
  The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The frequency and percentage of Grade 3+ adverse events will be reported.

OTHER OUTCOMES:
TOP1-deoxyribonucleic acid covalent complexes (TOP1cc) | Up to cycle 1 day 8 (1 cycle = 21 days)
  TOP1cc will be assessed on archival tissue and from pre-treatment and day 8 biopsies. The primary analysis is the relationship between induction of TOP1cc and individual responses. TOP1cc will be summarized for each sample as the percent of tumor cells with > 8 nucleoplasmic TOP1ccs. The change in TOP1cc from pre-treatment and day 8 samples (DTOP1cc) will be compared between responders and non-responders via two-sample t-tests. TOP1cc will be assessed in circulating tumor cells (CTC) from samples drawn pretreatment, cycle 1 day 2 and cycle 1 day 8. Presence of TOPcc in CTC will be examined graphically in an exploratory fashion. If feasible, comparisons of quantification between TOPcc in tissue versus CTC will be performed using Spearman correlation and scatter plots and association between TOPcc in CTC and response will be assessed as in tissue samples.
Homologous recombination (HR) status | Up to cycle 1 day 8 (1 cycle = 21 days)
  (HR) status (deficient versus proficient) will be assessed via staining for RAD51 foci on pretreatment and day 8 tumor biopsies. HR status will be compared to tumor response via chi-squared tests.
Protein expression | Up to cycle 1 day 8 (1 cycle = 21 days)
  Protein expression of ABCG2 will be measured via immunohistochemistry (IHC) on archival and pretreatment biopsies. H-scores will be used to score IHC staining, and H-scores will be compared between responders and non-responders using two-sample t-tests as indicated for TOP1cc.
Correlative analyses | Up to 5 years
  Exploratory analyses examining the association between correlative endpoints and other clinical endpoints (PFS and OS) may also be performed using Cox proportional hazards models and Kaplan Meier curves.
Gut microbiome analysis | Up to 5 years
  Data will be summarized by descriptive statistics, and non-parametric statistics and Principal Coordinate Analysis of Bray Curtis and weighted and unweighted UniFrac distances will be used to test for differences between cases with and without grade 3-4 diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea E. Wahner Hendrickson, M.D., Principal Investigator — Mayo Clinic in Rochester; Scott H. Kaufmann, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials